CLINICAL TRIAL: NCT03107637
Title: Therapeutic Implications of Early Transesophageal Echocardiography in Embolic Stroke of Undetermined Source (ESUS)
Brief Title: Transesophageal Echocardiography in Embolic Stroke of Undetermined Source
Acronym: ETO
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: NBS_2016_12
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Embolic Stroke of Undetermined Source; Ischemic Stroke
Keywords: Embolic Stroke of Undetermined Source; transesophageal echocardiography; cardiac source of embolism; ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
The ESUS concept was introduced recently to describe a non-lacunar stroke of undetermined etiology. The following etiological workup is required in this setting: head CT or MRI, 12-lead ECG, transthoracic echocardiography, continuous cardiac monitoring for at least 24 hours after stroke, vascular imaging (ultrasound, magnetic resonance angiography, CT angiography, catheter angiography). Transesophageal echocardiography (TEE) is considered not to be required.

However, aortic arch atheroma as diagnosed by TEE in the setting of recent ischemic stroke is a major aortic source of embolism, as supported by numerous well conducted studies. The European Association of Echocardiography considers that TEE is the gold standard for the diagnosis and the characterization of aortic atheroma. It is also the method of choice for the diagnosis of infectious endocarditis.

The aim of this work was to evaluate the rate of patients with a therapeutic modification induced by TEE (mainly anticoagulation and surgery), in consecutive patients admitted with ESUS at our institution stroke unit.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with a new onset of ischemic stroke
* Meeting the ESUS criteria (Embolic Stroke of Undetermined Source)
* Comprehensive transthoracic echo prior to the TEE

Exclusion Criteria:

* ESUS criteria not met
* Contraindications to TEE
* TEE failure
* Pregnant or breastfeeding woman
* Person under legal protection
* No medical insurance coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed for ichemic stroke meeting embolic source of unknown source criteria
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
therapeutic modification after transesophageal echocardiography | 24 hours after TEE
  proportion of patients with a therapeutic modification (mainly anticoagulation and surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Benyounes, MD, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (1):
- Fondation Ophtalmologique A de Rothschild, Paris, France